CLINICAL TRIAL: NCT01269710
Title: Second-Generation Antipsychotic Treatment Indication Effectiveness And Tolerability In Youth (Satiety) Study
Acronym: SATIETY
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Linmarie Sikich, MD, Associate Professor of Psychiatry, University of North Carolina, Chapel Hill
Other Study IDs: 09-1734
Record Dates: First submitted 2011-01-03; First posted 2011-01-04 (Estimated); Results first posted 2013-02-22 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-01

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorder; Psychotic Disorder, Not Otherwise Specified; Prodromal Schizophrenia; Mood Disorder; Bipolar Disorder; Major Depressive Disorder; Depressive Disorder, Not Otherwise Specified; Mood Disorder, Not Otherwise Specified; Autism Spectrum Disorder
Keywords: Second Generation Antipsychotics; Schizophrenia; Schizoaffective; Schizophreniform; Psychosis NOS; Mood Disorders; Weight; Autism
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Schizotypal Personality Disorder; Mood Disorders; Bipolar Disorder; Depressive Disorder, Major; Depressive Disorder; Autism Spectrum Disorder; Mental Disorders; Body Weight; Autistic Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — fasting glucose, lipid profile, insulin, leptin, prolactin, AST, ALT, CRP, adiponectin, ghrelin, cortisol, and relevant cytokines or peptide hormones (e.g., NP-Y, resistin, TNF-alpha, IL-1b, IL-2, IL-6, IL-8, IL-12, IL-18), sex hormones (e.g., testosterone, dehydroepiandrosterone, estrogen, luteinizing hormone, follicle stimulating hormone, and sex hormone binding globulin), and SGAP level (not baseline), to assure compliance. TSH and CBC will be measured at baseline only.
  Each subject will be asked to provide an additional 16 ml blood sample (approximately 1 tablespoon) for DNA collection and genotyping.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to get a better understanding of the side effect burden and identify predictors of psychotic, mood and aggressive disorders in children and adolescents. The study's primary aim is to identify genetic risk factors for weight gain and metabolic abnormalities.

DETAILED DESCRIPTION:
Participants will be evaluated for biological and genetic risk factors for nutritional and metabolic adverse effects associated with SGAPs (second generation antipsychotics) during 4 visits over 12 weeks. Participants will also be evaluated at month 6, 9, and 12. This study does not involve treatment for participants. Treatment of subjects enrolled in this study will be determined by their clinician and will remain unaffected by participation in this observational minimal risk study.

All participants were prescribed risperidone (Risperdal) for the duration of study participation and doses ranged from 0.25mg to 6mg daily for 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between the ages of 3 and 19 (at the time of consent)
2. Clinical diagnosis of psychotic disorders (i.e., schizophrenia, schizoaffective disorder, schizophreniform disorder, psychotic disorder not otherwise specified and prodromal schizophrenia (as defined by the Scale of Prodromal Symptoms (SOPS: Miller 1996)), mood disorder (i.e., bipolar disorder, major depressive disorder, depressive disorder not otherwise specified, mood disorder not otherwise specified) or an autism spectrum disorder.
3. Subjects who are considered for treatment with second generation antipsychotics (SGAPs) by a physician who has evaluated him/her
4. Subjects who are either A) antipsychotic naïve and have started an SGA within the past 2 weeks , B) have started a new antipsychotic within the past 2 weeks (specifically within 2 weeks of their first blood draw), or

Exclusion Criteria:

1. Individuals younger than 3 years or older than 19 years and 11 months (at the time of consent)
2. Personal history of or comorbid eating disorders
3. Active hyper-/hypothyroidism
4. Pregnancy
5. Severe medical disorder (i.e., AIDS, cancer, sepsis, etc.).

Ages: 3 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The investigators aim to recruit 200 individuals between the ages of 3 and 19, from a diverse range of ethnic and racial backgrounds, who have a clinical diagnosis of psychotic disorders, mood disorder or an autism spectrum disorder and are considered for treatment with second generation antipsychotic (SGAP) medication by a physician.
  Every effort will be made to recruit participants of all ethnicities, races and genders. The investigators will specifically target recruitment efforts toward minorities by using minority media and informational liaison with community organizations that serve minority populations.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2009-10; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects will be recruited from outpatient child psychiatry programs (including community clinics, school based mental health programs, private practices), inpatient psychiatry units and community outreach efforts.
Pre-assignment Details: Treatment of subjects enrolled in this study will be determined by their clinician and will remain unaffected by participation in this observational minimal risk study.
Groups:
- Observed Treatment Group: Participants in the observed treatment group will include up to 200 individuals between the ages of 3 and 19 who have a clinical diagnosis of psychotic spectrum, mood spectrum, or autism spectrum disorder and are considered for treatment with a second generation antipsychotic (SGA) by their treating clinician.
  Participants will be evaluated for biological and genetic risk factors for nutritional and metabolic adverse effects associated with SGAs during 4 visits over 12 weeks. Participants will also be evaluated at Month 6, 9, and 12.
  All participants were prescribed risperidone (Risperdal) for the duration of study participation and doses ranged from 0.25 mg to 6 mg daily for 52 weeks.
Period: Overall Study
Arm/Group | Observed Treatment Group
Started | 4
Week 12 | 3
Week 36 | 2
Completed | 1 (This refers to Week 52.)
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Observed Treatment Group
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight (in Lbs.)
Description: Participants will be evaluated for biological and genetic risk factors for nutritional and metabolic adverse effects associated with second-generation antipsychotics (SGA's) during 4 visits over 12 weeks. Participants will also be evaluated at Month 6, 9, and 12 (Week 52).
  Since only a single participant finished the study and had assessments through Week 52, we compiled the data from all subject endpoints (1 Week 12 visit, 2 Week 36 visits, and 1 Week 52 visit) and this is the data reported below.
Time Frame: Baseline and 52 Weeks
Population: All four enrolled study participants were included in this analysis.
Measure: Mean (Standard Deviation); unit: lbs.
Arm/Group | Observed Treatment Group
Number analyzed (Participants) | 4
lbs. | 24.9 (20.09)

2. Secondary Outcome: Change in Glucose Levels (mg/dL)
Description: as for outcome 1
Time Frame: Baseline and 52 Weeks
Population: All four enrolled study participants were included in this analysis.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Observed Treatment Group
Number analyzed (Participants) | 4
mg/dL | -2.25 (5.38)

3. Secondary Outcome: Change in Total Cholesterol (mg/dL)
Description: as for outcome 1
Time Frame: Baseline and 52 Weeks
Population: All four enrolled study participants were included in this analysis.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Observed Treatment Group
Number analyzed (Participants) | 4
mg/dL | -8.75 (12.61)

4. Secondary Outcome: Change in Triglycerides (mg/dL)
Description: as for outcome 1
Time Frame: Baseline and 52 Weeks
Population: All four enrolled study participants were included in this analysis.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Observed Treatment Group
Number analyzed (Participants) | 4
mg/dL | 18.75 (61.15)

5. Secondary Outcome: Change in LDL (mg/dL)
Description: as for outcome 1
Time Frame: Baseline and 52 Weeks
Population: All four enrolled study participants were included in this analysis.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Observed Treatment Group
Number analyzed (Participants) | 4
mg/dL | -6.25 (4.57)

ADVERSE EVENTS:
Arm/Group | Observed Treatment Group
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

LIMITATIONS AND CAVEATS:
This study only enrolled 4 subjects, thus, sample size was a significant limitation. Further, since only a single subject completed to Week 52, it is difficult to determine treatment indication effectiveness with second generation antipsychotics.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No